CLINICAL TRIAL: NCT00011986
Title: A Phase III Randomized Trial Of Paclitaxel And Carboplatin Versus Triplet Or Sequential Doublet Combinations In Patients With Epithelial Ovarian Or Primary Peritoneal Carcinoma
Brief Title: Combination Chemotherapy in Treating Patients With Stage III or Stage IV Ovarian Epithelial Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: SWOG Cancer Research Network (Network); Medical Research Council (Other Government); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0182; NCI-2012-02376 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-G0182; CDR0000068467; ISRCTN41636183; MRC-ICON5; ECOG-G0182; GOG-0182 (Other: Gynecologic Oncology Group); GOG-0182 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Results first posted 2016-04-19 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2016-03

CONDITIONS: Primary Peritoneal Carcinoma; Stage III Ovarian Cancer; Stage IV Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Taxes; Carboplatin; Gemcitabine; Topotecan; trioctyl phosphine oxide

ARMS (5):
- Arm I (Active Comparator): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment continues every 3 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- Arm II (Experimental): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 and gemcitabine IV over 30 minutes on days 1 and 8.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Gemcitabine Hydrochloride
- Arm III (Experimental): Patients receive chemotherapy as in arm I during courses 1-8 and doxorubicin HCl liposome IV over 1 hour on day 1 during courses 1, 3, 5, and 7. Treatment continues as in arm I.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Pegylated Liposomal Doxorubicin Hydrochloride
- Arm IV (Experimental): Patients receive topotecan IV over 30 minutes on days 1-3 and carboplatin IV over 30 minutes on day 3. Treatment continues every 3 weeks for 4 courses. Patients then receive 4 courses of arm I chemotherapy.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Topotecan Hydrochloride
- Arm V (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and carboplatin IV over 30 minutes on day 8. Treatment continues every 3 weeks for 4 courses. Patients then receive 4 courses of arm I chemotherapy. Patients with initial unresectable or suboptimal residual disease (more than 1 cm) may undergo interval cytoreductive surgery between courses 4 and 5 of chemotherapy.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Gemcitabine Hydrochloride; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; TAX
Drug: Carboplatin — Given IV
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdC; dFdCyd
  Arms: Arm II; Arm V
Drug: Pegylated Liposomal Doxorubicin Hydrochloride
  Other Names: doxorubicin HCl liposome; TLC D-99
  Arms: Arm III
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Hycamtin; SKF S-104864-A; TOPO
  Arms: Arm IV
Procedure: Therapeutic Conventional Surgery — Undergo surgery
  Arms: Arm V

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which combination chemotherapy regimen is most effective in treating ovarian epithelial cancer and peritoneal cancer. Randomized phase III trial to compare the effectiveness of various combination chemotherapy regimens in treating patients who have stage III or stage IV ovarian cancer or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Compare the efficacy of paclitaxel and carboplatin with or without gemcitabine, doxorubicin HCl liposome, or topotecan, in terms of overall and progression-free survival, in patients with stage III or IV ovarian epithelial or serous primary peritoneal carcinoma.

Determine the response rate in patients with measurable disease treated with these regimens.

Compare the toxic effects of these regimens in these patients. Compare the complications in patients treated with these regimens. Determine the dose-intensity and cumulative dose delivery for these regimens in these patients.

OUTLINE:

This is a randomized, multicenter study. Patients are stratified into 1 of 3 strata according to extent of residual disease and plans for interval cytoreductive surgery: Stratum A: Optimal (microscopic or macroscopic) residual disease without plans for surgery Stratum B: Suboptimal residual disease without plans for surgery Stratum C: Suboptimal residual disease with plans for surgeryPatients are randomized to 1 of 5 treatment arms. Arm I: Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment continues every 3 weeks for 8 courses in the absence of disease progression or unacceptable toxicity. Arm II: Patients receive chemotherapy as in arm I and gemcitabine IV over 30 minutes on days 1 and 8. Treatment continues as in arm I. Arm III: Patients receive chemotherapy as in arm I during courses 1-8 and doxorubicin HCl liposome IV over 1 hour on day 1 during courses 1, 3, 5, and 7. Treatment continues as in arm I. Arm IV: Patients receive topotecan IV over 30 minutes on days 1-3 and carboplatin IV over 30 minutes on day 3. Treatment continues every 3 weeks for 4 courses. Patients then receive 4 courses of arm I chemotherapy. Arm V: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and carboplatin IV over 30 minutes on day 8. Treatment continues every 3 weeks for 4 courses. Patients then receive 4 courses of arm I chemotherapy. Patients with initial unresectable or suboptimal residual disease (more than 1 cm) may undergo interval cytoreductive surgery between courses 4 and 5 of chemotherapy. Patients are followed every 3 months for 2 years and then every 6 months.

PROJECTED ACCRUAL: Approximately 4,000-5,000 patients (800-1,000 per treatment arm) will be accrued for this study within 3.5-5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage III or IV ovarian epithelial or serous primaryperitoneal carcinoma
* The following are ineligible:

  * Germ cell tumors
  * Sex cord-stromal tumors
  * Carcinosarcomas
  * Mixed Mullerian tumors or carcinosarcomas
  * Metastatic carcinomas from other sites to theovary
  * Low malignant potential tumors, including micropapillary serouscarcinomas
  * Mucinous primary peritoneal carcinoma
* Prior ovarian low malignant potential tumor (borderline carcinoma) that was surgically resected with subsequent development of invasive adenocarcinoma allowed if no prior chemotherapy
* Optimal (no greater than 1 cm) or suboptimal residual disease after initial surgery
* Prior breast cancer allowed provided the following are true:

  * Disease-free for more than 5 years
  * No prior cytotoxic chemotherapy for breast cancer
* Prior or concurrent primary endometrial cancer allowed if the following conditions are met:

  * Stage no greater than IB
  * Less than 3 mm invasion without vascular or lymphatic invasion
  * No poorly differentiated subtypes, including papillary serous, clear cell, or other FIGO grade 3 lesions
* Performance status - GOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2.5 times ULN
* No acute hepatitis
* Creatinine no greater than 1.5 times ULN
* No unstable angina
* No myocardial infarction within the past 6 months
* No evidence of abnormal cardiac conduction (e.g., bundle branch block, heart block) unless stable for the past 6 months
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No greater than grade 1 sensory or motor neuropathy
* No active infection that requires antibiotics
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No severe or ongoing gastrointestinal bleeding that requires blood product support
* See Disease Characteristics
* Prior chemotherapy for cancer involving the abdominal cavity or pelvis allowed provided the following are true:

  * More than 3 years since prior therapy
  * No evidence of recurrent disease
* No prior radiotherapy to any portion of the abdominal cavity or pelvis
* Prior radiotherapy for localized breast, head and neck, or skin cancer allowed provided the following are true:

  * More than 3 years since prior therapy
  * No evidence of recurrent disease
* See Disease Characteristics
* No more than 12 weeks since prior surgical resection

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4312 (Actual)
Dates: Start 2001-01; Primary Completion 2010-03 (Actual); Study Completion 2013-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bookman, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Praiss AM, Miller A, Smith J, Lichtman SM, Bookman M, Aghajanian C, Sabbatini P, Backes F, Cohn DE, Argenta P, Friedlander M, Goodheart MJ, Mutch DG, Gershenson DM, Tewari KS, Wenham RM, Wahner Hendrickson AE, Lee RB, Gray H, Secord AA, Van Le L, O'Cearbhaill RE. Carboplatin dosing in the treatment of ovarian cancer: An NRG oncology group study. Gynecol Oncol. 2023 Jul;174:213-223. doi: 10.1016/j.ygyno.2023.05.013. Epub 2023 May 23. PMID 37229879
- [Derived] Sia TY, Tew WP, Purdy C, Chi DS, Menzin AW, Lovecchio JL, Bookman MA, Cohn DE, Teoh DG, Friedlander M, Bender D, Mutch DG, Gershenson DM, Tewari KS, Wenham RM, Wahner Hendrickson AE, Lee RB, Gray HJ, Secord AA, Van Le L, Lichtman SM. The effect of older age on treatment outcomes in women with advanced ovarian cancer receiving chemotherapy: An NRG-Oncology/Gynecologic Oncology Group (GOG-0182-ICON5) ancillary study. Gynecol Oncol. 2023 Jun;173:130-137. doi: 10.1016/j.ygyno.2023.03.018. Epub 2023 May 4. PMID 37148580
- [Derived] Rose PG, Java JJ, Salani R, Geller MA, Secord AA, Tewari KS, Bender DP, Mutch DG, Friedlander ML, Van Le L, Method MW, Hamilton CA, Lee RB, Wenham RM, Guntupalli SR, Markman M, Muggia FM, Armstrong DK, Bookman MA, Burger RA, Copeland LJ. Nomogram for Predicting Individual Survival After Recurrence of Advanced-Stage, High-Grade Ovarian Carcinoma. Obstet Gynecol. 2019 Feb;133(2):245-254. doi: 10.1097/AOG.0000000000003086. PMID 30633128
- [Derived] Han MK, Tayob N, Murray S, Dransfield MT, Washko G, Scanlon PD, Criner GJ, Casaburi R, Connett J, Lazarus SC, Albert R, Woodruff P, Martinez FJ. Predictors of chronic obstructive pulmonary disease exacerbation reduction in response to daily azithromycin therapy. Am J Respir Crit Care Med. 2014 Jun 15;189(12):1503-8. doi: 10.1164/rccm.201402-0207OC. PMID 24779680
- [Derived] Nickles Fader A, Java J, Ueda S, Bristow RE, Armstrong DK, Bookman MA, Gershenson DM; Gynecologic Oncology Group (GOG)*. Survival in women with grade 1 serous ovarian carcinoma. Obstet Gynecol. 2013 Aug;122(2 Pt 1):225-232. doi: 10.1097/AOG.0b013e31829ce7ec. PMID 23969788

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Received began 1/29/2001 and ended 1/28/2003. This was an interventional trial involving patients enrolled from the United States (US), Canada, United Kingdom (UK), Italy, Australia, and New Zealand.
Pre-assignment Details: This study involved patients enrolled from two cooperative groups with the plan to combine data. 3882 patients were enrolled from one cooperative group and 430 from the other. This report includes those patients from both groups.
Groups:
- Carbo/Taxol: Carboplatin AUC 6 IV on day 1 plus Paclitaxel 175 mg/m2 IV on day 1 x 8 cycles
- Carbo/Taxol/Gemcitabine: Carboplatin AUC 5 IV on day 1 plus Paclitaxel 175 mg/m2 IV on day 1 x 8 cycles plus Gemcitabine 800 mg/m2/dIV on days 1 and 8 x 8 cycles
- Carbo/Taxol/Doxil: Carboplatin AUC 5 IV on day 1 plus Paclitaxel 175 mg/m2 IV on day 1 x 8 cycles plus Doxil 30 mg/m2 IV every other cycle on day 1 x 8 cycles
- Carbo/Topotecan - Carbo/Taxol: Topotecan 1.25 mg/m2/dIV days 1-3 plus Carboplatin AUC 5 IV on day 3 plus x 4 cycles followed by Carboplatin AUC 6 IV on day 1 plus Paclitaxel 175 mg/m2 IV on day 1 x 4 cycles
- Carbo/Gemcitabine - Carbo/Taxol: Gemcitabine 1000 mg/m2/dIV on days 1 and 8 plus Carboplatin AUC 6 IV on day 8 plus x 4 cycles followed by Carboplatin AUC 6 IV on day 1 plus Paclitaxel 175 mg/m2 IV on day 1 x 4 cycles
Period: Overall Study
Arm/Group | Carbo/Taxol | Carbo/Taxol/Gemcitabine | Carbo/Taxol/Doxil | Carbo/Topotecan - Carbo/Taxol | Carbo/Gemcitabine - Carbo/Taxol
Started | 864 | 864 | 862 | 861 | 861
Initiated Treatment | 862 | 860 | 854 | 846 | 851
Completed | 864 | 864 | 862 | 861 | 861
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbo/Taxol | Carbo/Taxol/Gemcitabine | Carbo/Taxol/Doxil | Carbo/Topotecan - Carbo/Taxol | Carbo/Gemcitabine - Carbo/Taxol | Total
Number analyzed (Participants) | 864 | 864 | 862 | 861 | 861 | 4312
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (11.1) | 58.8 (10.8) | 59.0 (11.1) | 58.2 (11.0) | 58.9 (10.7) | 58.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 864 | 864 | 862 | 861 | 861 | 4312
  Male | 0 | 0 | 0 | 0 | 0 | 0
International Federation of Gynecology and Obstetrics (FIGO) Stage [Number; unit: participants] — FIGO Staging Classification: 1985.
  Stage III: Tumor involving one or both ovaries with peritoneal implants outside the pelvis and/or positive retroperitoneal or inguinal nodes. Superficial liver metastasis equals Stage III. Tumor is limited to the true pelvis but with histologically verified malignant extensions to small bowel or omentum.
  Stage IV: Growth involving one or both ovaries with distant metastasis. If pleural effusion is present there must be positive cytologic test results to allot a case to Stage IV. Parenchymal liver metastasis equals Stage IV.
  participants
    Stage III:see description for details | 724 | 749 | 743 | 744 | 721 | 3681
    Stage IV:see description for details | 140 | 115 | 119 | 117 | 140 | 631
Primary Site of Disease [Number; unit: participants]
  Ovary | 748 | 752 | 737 | 752 | 751 | 3740
  Peritoneum | 116 | 112 | 125 | 109 | 110 | 572
Size of Residual Disease [Number; unit: participants]
  Microscopic only | 197 | 218 | 206 | 220 | 203 | 1044
  ≤ 1 cm gross disease | 404 | 384 | 405 | 358 | 398 | 1949
  > 1 cm gross disease | 263 | 262 | 251 | 283 | 260 | 1319

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Proportion of participants whose overall survival exceeded 5 years.
Time Frame: Up to 9 years
Population: All enrolled participants.
Measure: Number; unit: Proportion of participants
Arm/Group | Carbo/Taxol | Carbo/Taxol/Gemcitabine | Carbo/Taxol/Doxil | Carbo/Topotecan - Carbo/Taxol | Carbo/Gemcitabine - Carbo/Taxol
Number analyzed (Participants) | 864 | 864 | 862 | 861 | 861
Proportion of participants | 0.35 | 0.34 | 0.39 | 0.34 | 0.30

2. Primary Outcome: Progression-free Survival
Description: Median duration in months of progression free survival.
Time Frame: From the date of enrollment to first progression or death or last contact, if alive and progression free.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carbo/Taxol | Carbo/Taxol/Gemcitabine | Carbo/Taxol/Doxil | Carbo/Topotecan - Carbo/Taxol | Carbo/Gemcitabine - Carbo/Taxol
Number analyzed (Participants) | 864 | 864 | 862 | 861 | 861
months | 16.0 [14.9 to 17.2] | 16.3 [15.1 to 17.7] | 16.4 [15.3 to 17.5] | 15.4 [14.7 to 16.3] | 15.4 [14.6 to 16.4]

3. Secondary Outcome: Number of Participants With Observed Adverse Effects (Grade 3 and Above) Assessed by Common Toxicity Criteria Version 2.0
Time Frame: Up to 9 years
Population: Eligible and treated participants
Measure: Count of Participants; unit: Participants
Groups:
- Grade 3 and Above on ToxicityCarbo/Taxol: Carboplatin AUC 6 IV on day 1 plus Paclitaxel 175 mg/m2 IV on day 1 x 8 cycles
- Grade 3 and Above on Carbo/Taxol/Gemcitabine: Carboplatin AUC 5 IV on day 1 plus Paclitaxel 175 mg/m2 IV on day 1 x 8 cycles plus Gemcitabine 800 mg/m2/dIV on days 1 and 8 x 8 cycles
- Grade 3 and Above on Carbo/Taxol/Doxil: Carboplatin AUC 5 IV on day 1 plus Paclitaxel 175 mg/m2 IV on day 1 x 8 cycles plus Doxil 30 mg/m2 IV every other cycle on day 1 x 8 cycles
- Grade 3 and Above on Carbo/Topotecan - Carbo/Taxol: Topotecan 1.25 mg/m2/dIV days 1-3 plus Carboplatin AUC 5 IV on day 3 plus x 4 cycles followed by Carboplatin AUC 6 IV on day 1 plus Paclitaxel 175 mg/m2 IV on day 1 x 4 cycles
- Grade 3 and Above on Carbo/Gemcitabine - Carbo/Taxol: Gemcitabine 1000 mg/m2/dIV on days 1 and 8 plus Carboplatin AUC 6 IV on day 8 plus x 4 cycles followed by Carboplatin AUC 6 IV on day 1 plus Paclitaxel 175 mg/m2 IV on day 1 x 4 cycles
Arm/Group | Grade 3 and Above on ToxicityCarbo/Taxol | Grade 3 and Above on Carbo/Taxol/Gemcitabine | Grade 3 and Above on Carbo/Taxol/Doxil | Grade 3 and Above on Carbo/Topotecan - Carbo/Taxol | Grade 3 and Above on Carbo/Gemcitabine - Carbo/Taxol
Number analyzed (Participants) | 862 | 860 | 854 | 846 | 851
Participants
  Leukopenia | 438 | 686 | 595 | 476 | 513
  Neutropenia | 749 | 798 | 782 | 779 | 761
  Thrombocytopenia | 193 | 520 | 320 | 303 | 486
  Anemia | 102 | 196 | 160 | 167 | 203
  Other Hematologic | 156 | 338 | 244 | 246 | 315
  Allergy | 38 | 20 | 28 | 21 | 26
  Auditory | 5 | 2 | 3 | 2 | 1
  Cardiovascular | 20 | 36 | 34 | 17 | 23
  Coagulation | 5 | 10 | 4 | 9 | 7
  Constitutional | 54 | 96 | 84 | 73 | 57
  Dermatologic | 13 | 6 | 11 | 6 | 8
  Endocrine | 0 | 4 | 2 | 1 | 1
  Gastrointestinal | 90 | 145 | 124 | 105 | 92
  Genitourinary/Renal | 9 | 8 | 13 | 6 | 9
  Hemorrhage | 8 | 29 | 20 | 8 | 30
  Hepatic | 13 | 32 | 11 | 13 | 25
  Infection/Fever | 76 | 138 | 134 | 84 | 82
  Metabolic | 61 | 55 | 55 | 37 | 45
  Musculoskeletal | 7 | 18 | 13 | 8 | 10
  Neurologic | 34 | 47 | 43 | 28 | 35
  Peripheral Neurologic | 45 | 59 | 45 | 35 | 24
  Ocular/Visual | 1 | 3 | 1 | 3 | 3
  Pain | 53 | 75 | 75 | 66 | 52
  Pulmonary | 19 | 37 | 39 | 21 | 37
  Sexual | 0 | 0 | 1 | 1 | 0
  Second Primary | 34 | 66 | 51 | 41 | 57

ADVERSE EVENTS:
Time Frame: From date of enrollment onto the study to 30 days after last treatment cycle or any Adverse Event (AE) considered to be due to study treatment regardless of when it occurred.
Description: Only Serious Adverse Events(SAE) for the US-enrolled participants is able to be reported. Due to the methods in which AEs were collected &/or stored, it is not possible to report only the Other(not including Serious) AEs in the appropriate table. Therefore that table is a combined set of SAEs & non-serious AEs. Other AEs are Grade 2 or worse.
Arm/Group | Carbo/Taxol | Carbo/Taxol/Gemcitabine | Carbo/Taxol/Doxil | Carbo/Topotecan - Carbo/Taxol | Carbo/Gemcitabine - Carbo/Taxol
Serious Adverse Events (participants affected / at risk) | 86/777 | 107/774 | 115/767 | 77/766 | 100/767
Other Adverse Events (participants affected / at risk) | 857/862 | 856/860 | 852/854 | 843/846 | 849/851
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carbo/Taxol (N=777) | Carbo/Taxol/Gemcitabine (N=774) | Carbo/Taxol/Doxil (N=767) | Carbo/Topotecan - Carbo/Taxol (N=766) | Carbo/Gemcitabine - Carbo/Taxol (N=767)
Allergy-Other (Immune system disorders) | 4 | 0 | 2 | 1 | 0
Allergic Reaction/Hypersensitivity (Immune system disorders) | 9 | 6 | 6 | 3 | 6
Inner Ear/Hearing (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Hearing-Other (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 2 | 2 | 1 | 0 | 3
Platelets (Blood and lymphatic system disorders) | 1 | 12 | 2 | 0 | 8
Neutrophils/Granulocytes (Blood and lymphatic system disorders) | 1 | 3 | 3 | 3 | 1
Leukocytes (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Cardiac disorders) | 1 | 0 | 0 | 1 | 1
Circulatory Or Cardiac-Other (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Cardiac Left Ventricular Function (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Cardiac Troponin I (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 2 | 0 | 0
Phlebitis (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Vasovagal Episode (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Supraventricular Arrhythmias (Cardiac disorders) | 1 | 1 | 1 | 0 | 1
Thrombosis/Embolism (Cardiac disorders) | 10 | 9 | 13 | 13 | 16
Nodal/Junctional Arrhythmia/Dysrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Arrhythmia- Other (Cardiac disorders) | 0 | 0 | 1 | 0 | 2
Cardiac-Ischemia/Infarction (Cardiac disorders) | 1 | 1 | 2 | 1 | 0
Sinus Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Edema (Cardiac disorders) | 0 | 1 | 0 | 1 | 1
Constitutional Symptoms-Other (General disorders) | 1 | 0 | 0 | 0 | 0
Fever In The Absence Of Neutropenia (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 3 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Wound-Infectious (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 2
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2
Skin-Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Wound-Non-Infectious (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Stomatitis/Pharyngitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gi-Other (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 5 | 4 | 2 | 4 | 5
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Anorexia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspepsia/Heartburn (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Ascites (Non-Malignant) (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1
Fistula-Rectal/Anal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Gastrointestinal disorders) | 2 | 3 | 2 | 2 | 1
Constipation (Gastrointestinal disorders) | 6 | 7 | 3 | 5 | 3
Diarrhea (Without Colostomy) (Gastrointestinal disorders) | 1 | 4 | 3 | 1 | 2
Vomiting (Gastrointestinal disorders) | 7 | 8 | 11 | 7 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1
Hemorrhage-Other (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Rectal Bleeding/Hematochezia (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Hemorrhage/Bleeding Associated With Surgery (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Hemorrhage/Bleeding With Grade 3 Or 4 Th (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hematuria (In The Absence Of Vaginal Bleeding (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hepatic-Other (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Sgpt (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Sgot (Hepatobiliary disorders) | 0 | 2 | 0 | 1 | 1
Bilirubin (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Infection, Other (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Catheter-Related Infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Infection With Unknown Anc (Infections and infestations) | 0 | 1 | 1 | 1 | 2
Infection Documented W Grd 3/4 Neutropn. (Infections and infestations) | 5 | 9 | 15 | 7 | 4
Infection Without Neutropenia (Infections and infestations) | 7 | 8 | 5 | 6 | 6
Febrile Neutropenia-Fuo Infect Not Docum (Infections and infestations) | 8 | 12 | 15 | 10 | 7
Metabolic-Other (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Hypomagnesmia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Joint, Muscle, Or Bone-Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Speech Impairment- Dysphasia/Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Seizure(S) (Nervous system disorders) | 1 | 0 | 0 | 0 | 2
Hallucinations (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cns Cerebrovascular Ischemia (Nervous system disorders) | 0 | 0 | 4 | 0 | 2
Confusion (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Syncope (Nervous system disorders) | 6 | 2 | 5 | 0 | 3
Mood Alteration-Anxiety Agitation (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Dizziness/Lightheadedness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Neuropathy-Sensory (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Neuropathy Motor (Nervous system disorders) | 1 | 1 | 1 | 0 | 1
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 0
Chest Pain Non-Cardiac Or Non-Pleuritic (General disorders) | 0 | 0 | 1 | 1 | 0
Headache (General disorders) | 0 | 0 | 1 | 0 | 0
Abdominal Pain Or Cramping (General disorders) | 4 | 3 | 4 | 1 | 1
Bone Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (General disorders) | 0 | 0 | 1 | 0 | 0
Myalgia (General disorders) | 1 | 0 | 0 | 0 | 0
Pain-Other (General disorders) | 0 | 1 | 1 | 0 | 1
Pleural Effusion (Non-Malignant) (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4 | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Operative Injury To Bladder/Ureter (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Fistula Or Gu Fistula (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 1
Creatinine (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Renal/Gu-Other (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Carbo/Taxol (N=862) | Carbo/Taxol/Gemcitabine (N=860) | Carbo/Taxol/Doxil (N=854) | Carbo/Topotecan - Carbo/Taxol (N=846) | Carbo/Gemcitabine - Carbo/Taxol (N=851)
Leukopenia (Blood and lymphatic system disorders) | 746 | 826 | 806 | 782 | 800
Neutropenia (Blood and lymphatic system disorders) | 821 | 838 | 818 | 830 | 825
Thrombocytopenia (Blood and lymphatic system disorders) | 319 | 675 | 438 | 460 | 645
Anemia (Blood and lymphatic system disorders) | 508 | 700 | 603 | 647 | 685
Other Hemotologic (Blood and lymphatic system disorders) | 164 | 351 | 261 | 260 | 327
Allergy (Immune system disorders) | 65 | 42 | 54 | 39 | 47
Auditory (Ear and labyrinth disorders) | 22 | 20 | 23 | 17 | 15
Cardiovascular (Cardiac disorders) | 43 | 72 | 62 | 36 | 61
Coagulation (Vascular disorders) | 10 | 12 | 6 | 14 | 10
Constitutional (General disorders) | 365 | 434 | 403 | 367 | 363
Dermatologic (Skin and subcutaneous tissue disorders) | 63 | 61 | 109 | 47 | 64
Endocrine (Endocrine disorders) | 36 | 38 | 41 | 40 | 27
Gastrointestinal (Gastrointestinal disorders) | 421 | 469 | 496 | 403 | 399
Genitourinary/Renal (Renal and urinary disorders) | 46 | 53 | 56 | 36 | 42
Hemorrhage (Blood and lymphatic system disorders) | 14 | 41 | 33 | 18 | 50
Hepatic (Hepatobiliary disorders) | 43 | 96 | 42 | 39 | 79
Infection/Fever (Infections and infestations) | 135 | 196 | 199 | 143 | 147
Metabolic (Metabolism and nutrition disorders) | 118 | 98 | 107 | 79 | 97
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 55 | 62 | 52 | 44 | 45
Neurologic (Nervous system disorders) | 117 | 135 | 110 | 90 | 119
Peripheral neurologic (Nervous system disorders) | 207 | 232 | 207 | 134 | 144
Ocular/Visual (Eye disorders) | 42 | 54 | 64 | 28 | 38
Pain (General disorders) | 317 | 301 | 294 | 295 | 289
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 104/861 | 129 | 118 | 106 | 145
Sexual (Reproductive system and breast disorders) | 4 | 9 | 11 | 6 | 5
2nd Primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 70 | 94 | 85 | 74 | 85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No